CLINICAL TRIAL: NCT06209489
Title: The Effect of White Cover and Massage Application on Bilirubin Level and Duration of Phototherapy in Newborns Undergoing Phototherapy
Brief Title: White Cover and Massage Impact on Bilirubin Levels and Phototherapy Duration in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Zeynep ÇİFTCİ DEMİRTAŞ, Midwife, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-77192459-050.99-299327
Record Dates: First submitted 2023-12-30; First posted 2024-01-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Newborn Jaundice; Hyperbilirubinemia, Neonatal; Newborn Massage; Phototerapy; White Cover
Keywords: Newborn; Phototherapy; White Cover; Massage; Hyperbilirubinemia
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): 1. White fabric will be covered over the incubator for term newborns during phototherapy.
  2. During phototherapy, term newborns will receive a baby massage, including facial massage, chest massage, arm massage, abdominal massage and leg massage, twice a day for 15 minutes.
  Interventions: Other: White cover
- Control group (No Intervention): The hospital's clinical routine will be applied to the newborns in the control group.

INTERVENTIONS:
Other: White cover — * A white cover will be covered over the incubator during phototherapy.
  * Baby massage will be applied during phototherapy.
  Other Names: Newborn massage
  Arms: İntervention group

SUMMARY:
This study aimed to examine the effect of white cover and massage application on newborns' bilirubin level and duration of phototherapy in newborns receiving phototherapy.

DETAILED DESCRIPTION:
Hyperbilirubinemia is a common problem seen in the neonatal period, characterized by yellow staining of the skin and sclera, causing an increase in total serum bilirubin >5 mg/dl. Neonatal jaundice is seen in 60% of term newborns and 80% of preterm newborns. Hyperbilirubinemia is usually physiological and disappears within a few days. Jaundice may worsen and lead to kernicterus (accumulation of bilirubin in some parts of the brain) or death if pathological hyperbilirubinemia occurs. Therefore, every baby with hyperbilirubinemia and high serum bilirubin levels requires serious attention and treatment. The primary treatment for neonatal jaundice is phototherapy. The effectiveness of phototherapy depends on the phototherapy light source, light intensity, distance between the phototherapy light and the newborn, and the body surface area exposed to the light. Phototherapy has potential side effects in newborns such as hyperthermia, dehydration, diarrhea, bronze baby syndrome, and skin burns. For this reason, the use of phototherapy should be minimized and solutions should be found to shorten the duration of phototherapy. To increase the effectiveness of phototherapy treatment, a reflector material can be added to the phototherapy. White fabric, which can be used as a reflector, can reflect scattered phototherapy light. When fabrics made of reflective materials are hung over the phototherapy device, they can capture the light that may scatter from the baby to the environment and reflect the light back to the baby. White fabric may increase irradiance and therefore lead to increased bilirubin conversion.Studies have reported that massage applied before phototherapy is effective in reducing the bilirubin level in babies with hyperbilirubinemia. Bilirubin is eliminated from the body through defecation. Removing bilirubin from the body reduces jaundice. Massage reduces bilirubin levels by increasing the frequency of bowel movements in newborn babies.

ELIGIBILITY:
Inclusion Criteria:

* Term babies with gestational age between 37-42 weeks,
* Does not have a respiratory, cardiovascular, gastrointestinal or neurological disorder or syndrome that would prevent or complicate oral feeding,
* Birth weight of 2500 g and above,
* With phototherapy indication,
* Do not have any health problems other than neonatal jaundice detected in the prenatal period,
* Those with a stable health condition,
* Orally fed,
* No clinical signs of dehydration,
* Do not have any skin problems that would prevent baby massage,
* Newborns with written and verbal informed consent from their families will be included in the study.

Exclusion Criteria:

* Premature,
* Those with congenital malformations,
* Those with hyperbilirubinemia requiring exchange transfusion,
* Those with Rh hemolytic disease,
* Having a positive culture test (sepsis),
* Those with glucose-6-phosphate dehydrogenase (G6PD) deficiency,
* Birth weight below 2500 grams,
* Those who were referred to another center during the research,
* Discharged early,
* Unexpected complications developed during the research,
* Bronze child syndrome occurs during phototherapy,
* Newborns who develop a pathology that will prevent or complicate oral feeding will not be included in the study.

Ages: 12 Hours to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
White cover | 24 hours
  A white cover will be covered over the incubator during phototherapy.
Newborn massage | 2 times 15 minutes at 12 hour intervals
  Baby massage will be applied during phototherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep ZE ÇİFTCİ DEMİRTAŞ, 1, Principal Investigator — midwife
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No